CLINICAL TRIAL: NCT07010926
Title: A Double-Blind, Randomized, Placebo-Controlled Phase II Clinical Trial to Evaluate the Safety and Efficacy of L2-01 in Subjects With Crohn's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: L2 Bio, LLC (Industry)
Collaborators: FDAMap (Unknown); Akan Biosciences, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L2-01-CD
Record Dates: First submitted 2025-05-29; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Crohn&Amp;#39;s; Crohn&Amp;#39;s Disease (CD)
Keywords: Crohn's Disease; Stem Cells; Autologous; Mesenchymal Stem Cells (MSC); Adipose; Crohn's

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study monitors will also be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L2-01 Treatment Arm (Experimental): Participants in this arm receive a single intravenous infusion of L2-01, a human adipose-derived mesenchymal stem cell product. The dose is 1 × 10^6 MSC cells per kilogram of body weight, suspended in 10 ml of lactated Ringer's solution mixed with 100 ml of saline. The infusion is administered over approximately 30 minutes. MSCs are derived from the patient's own adipose tissue or from that of a first-degree relative.
  Interventions: Biological: L2-01 adipose-derived mesenchymal stem cells (MSC)
- Placebo Comparator Arm (Placebo Comparator): Participants in this arm receive a single intravenous infusion of placebo, consisting of 10 ml of lactated Ringer's solution mixed with 100 ml of saline. The infusion is administered over approximately 30 minutes. The placebo product is packaged identically to the active product to maintain study blinding.
  Interventions: Other: Placebo saline solution

INTERVENTIONS:
Biological: L2-01 adipose-derived mesenchymal stem cells (MSC) — L2-01 is a biological product consisting of human mesenchymal stem cells isolated from adipose tissue of the patient or a first-degree relative. The MSCs are expanded under Good Manufacturing Practice (GMP) conditions and suspended in 10 ml of lactated Ringer's solution. The product is administered as a single intravenous infusion at a dose of 1 × 10^6 cells per kilogram of body weight, diluted in 100 ml of saline, infused over approximately 30 minutes. The infusion is closely monitored for safety.
  Arms: L2-01 Treatment Arm
Other: Placebo saline solution — Placebo consists of 10 ml of lactated Ringer's solution mixed with 100 ml of saline. It is administered as a single intravenous infusion over approximately 30 minutes. The placebo is packaged identically to the active product to maintain study blinding.
  Arms: Placebo Comparator Arm

SUMMARY:
This clinical trial is testing a new treatment called L2-01 in patients with Crohn's Disease, a condition that causes ongoing inflammation of the digestive tract. Current treatments for Crohn's Disease do not work for everyone, and some patients still experience symptoms even with standard therapies.

The purpose of this study is to determine if a single intravenous infusion of L2-01, which uses cells called mesenchymal stem cells derived from a patient's own or their close relative's body fat, is safe and can help improve symptoms of Crohn's Disease. Researchers will compare the effects of L2-01 to a placebo (an inactive substance) to see if L2-01 helps reduce inflammation and improves quality of life in patients.

The main questions the study aims to answer are:

Is L2-01 safe for patients with Crohn's Disease?

Can L2-01 effectively reduce symptoms and improve the health of people living with Crohn's Disease compared to a placebo?

The researchers believe that L2-01 will be safe and more effective than placebo in reducing inflammation, decreasing disease activity, and improving patients' quality of life.

DETAILED DESCRIPTION:
This Phase II clinical trial is a randomized, double-blind, placebo-controlled study designed to evaluate the safety and efficacy of L2-01, a human adipose-derived mesenchymal stem cell (MSC) product, in patients with Crohn's Disease (CD). L2-01 consists of MSCs harvested from the patient's own adipose tissue or that of a first-degree relative, expanded in culture, and administered as a single intravenous infusion at a dose of 1 × 10^6 cells per kilogram of body weight.

The study enrolls 120 adult subjects with non-active Crohn's Disease, defined by a Crohn's Disease Activity Index (CDAI) of 200 or less. Patients are randomized in a 1:1 ratio to receive either L2-01 or placebo (sterile normal saline). The initial 20 patients are enrolled in a staggered manner to closely monitor safety signals, followed by enrollment of an additional 100 subjects if no significant adverse drug reactions are observed.

Subjects undergo liposuction to collect approximately 25 ml of lipoaspirate from the lower abdomen or flanks under local anesthesia. The MSCs are isolated, expanded under Good Manufacturing Practice (GMP) conditions, cryopreserved, and then thawed and prepared as a ready-to-infuse suspension prior to administration. Placebo infusions contain an identical volume of lactated Ringer's solution mixed with saline, maintaining blinding integrity.

The infusion is administered intravenously over approximately 30 minutes with close monitoring for adverse events, vital sign changes, and infusion reactions during and after the procedure. Safety assessments include monitoring treatment-emergent adverse events (TEAEs), laboratory tests (including comprehensive metabolic panel, complete blood count, coagulation studies, and inflammatory markers), physical examinations, vital signs, and adverse event reporting per MedDRA coding.

Efficacy assessments focus on changes in systemic disease activity, inflammatory markers, imaging (pelvic MRI), and quality of life metrics (using the IBDQ-32 questionnaire). Follow-up visits occur at scheduled intervals up to 24 weeks post-infusion to assess both safety and therapeutic effects.

Quality assurance for the study includes routine source data verification by the Contract Research Organization (CRO) monitors, adherence to International Council for Harmonisation (ICH) Good Clinical Practice (GCP) guidelines, and oversight by an independent Data Safety Monitoring Board (DSMB) composed of physicians and regulatory experts who review safety data in real time. Investigational product handling, storage, and accountability procedures are strictly controlled and documented.

Statistical analyses are primarily descriptive with 95% confidence intervals, focusing on safety endpoints in the intent-to-treat (ITT) population. No formal interim analyses are planned; however, stopping rules are predefined for severe adverse events or safety concerns related to the investigational product or procedures. The study aims to provide clinically meaningful data to support further development of L2-01 as a novel immunomodulatory therapy for Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Crohn Disease (CD) diagnosed within 12 months before acceptance of clinical, endoscopical, anatomopathological and/or radiological criteria and have a non-active CD. (Crohn´s Disease Activity Index (CDAI)≤ 200)
2. Any gender, > 18 Years of age
3. Negative pregnancy test in female subjects
4. Patients voluntarily sign the informed consent before performance of any study-related procedures
5. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements

Exclusion Criteria:

1. Patients who have received infliximab or any other anti-TNF agent within 8 weeks before the cell treatment administration.
2. Patients who have received tacrolimus or cyclosporine within 4 weeks before cell treatment.
3. Patients with a history of alcohol or other addictive substance abuse within 6 months before inclusion.
4. Severe uncontrolled diseases (chronic renal failure, cardio, pulmonary, etc.).
5. Any type of medical or psychiatric disease which are considered an exclusion criterion, in the investigator's opinion.
6. Patients with a diagnosis of malignant neoplasia, except basal cell or epidermoid carcinoma of the skin, or a previous history of malignant tumors, except those that have no evidence of relapse for at least 5 years.
7. Subjects with congenital or acquired immunodeficiency.
8. Subjects who tested positive for HIV 1/2, HBV, HCV, HTLV I/II, WNV, and syphilis
9. Flu symptoms
10. Patient had major surgery or serious trauma within 6 weeks before enrolment.
11. Pregnant or breastfeeding women.
12. Physical or psychological impossibility of following the protocol requirements
13. Patients who are receiving or have received another investigational drug within 30 days prior to the first visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events occurring in less than 5% of study participants as a measure of safety. | From the day of infusion through 12 weeks post-infusion.

SECONDARY OUTCOMES:
Change in Crohn's Disease Activity Index (CDAI) from baseline to 12 weeks post-infusion. | Baseline and 12 weeks post-infusion.
Improvement in inflammatory markers and MRI results from baseline to 12 weeks post-infusion. | Baseline and 12 weeks post-infusion.
Change in quality of life as assessed by the Inflammatory Bowel Disease Questionnaire (IBDQ-32) from baseline to 12 weeks post-infusion. | Baseline and 12 weeks post-infusion.
Relapse rate among patients who achieved treatment success with adipose-derived mesenchymal stem cells. | Up to 24 weeks post-infusion.
Biological characterization of the cell product (phenotype study, suppressor capacity, cytokine production) and its correlation with therapeutic effect. | At infusion and during follow-up assessments up to 24 weeks.

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), withdrawals due to adverse events, changes in laboratory values, and vital signs. | From day of infusion through 24 weeks post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Kumar, PhD, RAC, Study Director — FDAMap

IPD SHARING:
Plan to Share IPD: Undecided